CLINICAL TRIAL: NCT05636059
Title: Comparative Effects of Different Physiotherapy Methods on Pain, Function and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Physiotherapy in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LithuanianSportsU-12
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee function; womac; quality of life; joint mobilization; physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy; Exercise; Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Experimental): 32 sessions in total, 2 times a day, 30 min. one session. Exercise program consisted of: cycling stationary bike, isometric and isotonic exercise for knee flexion / extension, hip flexion / extension / abduction / adduction, exercise with resistance bands, weights, and gymnastic ball.
  Interventions: Other: Therapeutic exercise
- Exercise + cryotherapy (Experimental): Exercise program - 16 sessions in total, once a day, 30 min. one session. Cryotherapy - 8 sessions in total, two-three times a week, one session - 2 min. duration, temperature -60 to -140 C degrees.
  Exercise program consisted of: cycling stationary bike, isometric and isotonic exercise for knee flexion / extension, hip flexion / extension / abduction / adduction, exercise with resistance bands, weights, and gymnastic ball.
  Interventions: Other: Exercise + cryotherapy
- Exercise + joint mobilization (Experimental): Exercise program - 16 sessions in total, once a day, 30 min. one session, two-three times a week.
  Joint mobilization - 8 sessions in total, anterior - posterior tibia femoral glide, patella motion, lateral and medial movement.
  Exercise program consisted of: cycling stationary bike, isometric and isotonic exercise for knee flexion / extension, hip flexion / extension / abduction / adduction, exercise with resistance bands, weights, and gymnastic ball.
  Interventions: Other: Exercise + joint mobilization

INTERVENTIONS:
Other: Therapeutic exercise — 32 sessions in total, 2 times a day, 30 min. one session. Exercise program consisted of: cycling stationary bike, isometric and isotonic exercise for knee flexion / extension, hip flexion / extension / abduction / adduction, exercise with resistance bands, weights, and gymnastic ball.
  Arms: Exercise
Other: Exercise + cryotherapy — Exercise program - 16 sessions in total, once a day, 30 min. one session. Cryotherapy - 8 sessions in total, two-three times a week, one session - 2 min. duration, temperature -60 to -140 C degrees.
  Exercise program consisted of: cycling stationary bike, isometric and isotonic exercise for knee flexion / extension, hip flexion / extension / abduction / adduction, exercise with resistance bands, weights, and gymnastic ball.
  Arms: Exercise + cryotherapy
Other: Exercise + joint mobilization — Exercise program - 16 sessions in total, once a day, 30 min. one session, two-three times a week.
  Joint mobilization - 8 sessions in total, anterior - posterior tibia femoral glide, patella motion, lateral and medial movement.
  Exercise program consisted of: cycling stationary bike, isometric and isotonic exercise for knee flexion / extension, hip flexion / extension / abduction / adduction, exercise with resistance bands, weights, and gymnastic ball.
  Arms: Exercise + joint mobilization

SUMMARY:
Osteoarthritis symptoms can be managed with non-drug treatments such as patient education, exercise or weight loss interventions. Cryotherapy is one of the effective method to reduce joint inflammation, pain and improve function. Another method is joint mobilization, which can also reduce pain and improve function. Based on this theory, it was hypothesized that cryotherapy will have better effect on pain and the quality of life, whereas joint mobilization will be more effective on knee function. The aim of the study was to compare the effects of different physiotherapy methods on pain, knee joint function and quality of life in individuals with osteoarthritis.

DETAILED DESCRIPTION:
Study included 63 participants with knee osteoarthritis. All subjects were randomly assigned to one of 3 groups: exercise group (n=21), exercise + cryotherapy group (n=21), or exercise + joint mobilization group (n=21). VAS scale was used to assess the pain, quality of life was evaluated with Short Form 36 Health Survey Questionnaire (SF-36) questionnaire, knee ranges of motion were measured using a goniometer, strength of the muscles was assessed on the Oxford 5 point scale, The Western Ontario and McMaster Universities Arthritis Index (WOMAC) was used to evaluate knee osteoarthritis. All the participants received 30 intervention sessions.

ELIGIBILITY:
Inclusion Criteria:

* stage II of the knee OA;
* affected knee joint;
* pain of at least 3 points on the VAS.

Exclusion Criteria:

* Severe cardiovascular disease;
* Oncological Disorders;
* Allergy to cold / cold intolerance;
* Impaired lower limbs blood circulation;
* Fear of confined spaces;
* Pregnancy or lactation.

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain at 18 days | Baseline and after 18 days
  Pain was assessed using a visual analogue scale (VAS) that used a 10-cm line with end-point descriptors such as 'no pain' marked at the left end and 'worst pain imaginable' marked at the right end. Patients were asked to mark a point on the line that best represented their pain at the time of the evaluation. The distance from 'no pain' to the patient's mark was then measured and recorded as the VAS score: 0 cm was defined as no pain, 1-3 cm as mild pain, 4 or 5 cm as moderate pain, 6-8 cm as severe pain and 9 or 10 cm as the worst pain imaginable.
Change from baseline Quality of Life at 18 days | Baseline and after 18 days
  The SF-36 quality of life questionnaire is used to assess health-related quality of life. The questionnaire consists of 36 questions and reflects 8 areas of life: physical activity, activity limitation due to physical ailments and/or emotional disorders, social relationships, emotional state, energy and vitality, pain, general health assessment. The questionnaire can be completed by the subject or by a specialist conducting the study. Answers are scored. Numerical value of each area from 0 to 100 points. The more points collected, the better the quality of life. Test reliability is 0.791.
Change from baseline Knee Ranges of Motions at 18 days | Baseline and after 18 days
  Using goniometer the range of knee motions were evaluated: flexion, extension. Each motion was measured three times and averaged value was used.
Change from baseline Knee Muscle Strength at 18 days | Baseline and after 18 days
  The muscle strength of knee flexion and extension was evaluated using manual muscle testing technique (Oxford 5 point scale).
Change from baseline Knee Health Status at 18 days | Baseline and after 18 days
  Self-administered Western Ontario and McMaster Universities (WOMAC) index was used to to quantify the health status of patients with knee osteoarthritis. It is the most common used clinical tools for evaluating patients with knee OA. It includes five questions about pain, two about stiffness, and 17 on degree of disability of activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Dudonienė, PhD, Study Director — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

REFERENCES:
- [Derived] Dudoniene V, Bitinas D, Zlibinaite L. Comparison of three different therapeutic interventions in the management of knee osteoarthritis: Randomized controlled parallel group pilot trial. Osteoarthr Cartil Open. 2025 Oct 17;7(4):100697. doi: 10.1016/j.ocarto.2025.100697. eCollection 2025 Dec. PMID 41211535